CLINICAL TRIAL: NCT03165799
Title: Mindfulness to the Clinical Setting: The Mind Hand Connection Study
Acronym: MHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vineet Chopra, Chief, Division of Hospital Medicine & Assistant Professor of Medicine & Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-020159-0004
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Mindfulness; Education, Medical; Hand Hygiene; Patient Safety

STUDY DESIGN:
Intervention Model Description: Participating teams were randomized with a 1:1 ratio to receive the intervention.
Who Masked: Outcomes Assessor
Masking Description: Observers collecting data were blinded to participant treatment/control randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Education (Experimental): Participants viewed an informational video titled, "All it Takes is 10 Mindful Minutes" by mindfulness expert, Andy Puddicombe. Following the video, a guided discussion was provided that focused on how the principles of mindfulness can be used to influence a physician's state of mental presence, allowing for moments of clarity, insight, and reflection, and potentially enhance provider and patient safety.
  Interventions: Behavioral: Mindfulness Education
- No Intervention (No Intervention): Participants did not receive mindfulness education.

INTERVENTIONS:
Behavioral: Mindfulness Education — Mindfulness Education
  Arms: Mindfulness Education

SUMMARY:
This is a single center, randomized study that assessed the effects of mindfulness training on physician teaching teams at a VA hospital.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate changes in hand hygiene compliance pre- and post- intervention in Internal Medicine physician and medical student inpatient teaching teams. Half of the teaching teams received the intervention of mindfulness education. Blinded observers collected data on hand hygiene compliance and mindfulness behaviors for both teams during patient care rounds for 1-week pre and post intervention. Additionally, the intervention group participated in focus group/interview discussions.

ELIGIBILITY:
Inclusion Criteria:

Internal Medicine attendings, residents, interns and medical students on inpatient patient care teams, able to provide consent

Exclusion Criteria:

Surgical attendings, residents, interns or subspeciality teams, Internal medicine attendings rotating on non-resident teams

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Hand Hygiene Compliance | Baseline and study completion at 2 weeks
  Change in hand hygiene compliance observed during patient care rounds

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale | Baseline and study completion at 2 weeks
  Measures core characteristics of mindfulness

CONTACTS AND LOCATIONS:
Overall Officials: Vineet I Chopra, MD, Principal Investigator — University of Michigan and Ann Arbor VA Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilmartin HM. Use hand cleaning to prompt mindfulness in clinic. BMJ. 2016 Jan 4;352:i13. doi: 10.1136/bmj.i13. No abstract available. PMID 26728590
- [Background] Kiyoshi-Teo H, Krein SL, Saint S. Applying mindful evidence-based practice at the bedside: using catheter-associated urinary tract infection as a model. Infect Control Hosp Epidemiol. 2013 Oct;34(10):1099-101. doi: 10.1086/673147. Epub 2013 Aug 23. PMID 24018928
- [Background] Ellingson K, Haas JP, Aiello AE, Kusek L, Maragakis LL, Olmsted RN, Perencevich E, Polgreen PM, Schweizer ML, Trexler P, VanAmringe M, Yokoe DS. Strategies to prevent healthcare-associated infections through hand hygiene. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S155-78. doi: 10.1017/s0899823x00193900. No abstract available. PMID 25376074
- [Background] King D, Vlaev I, Everett-Thomas R, Fitzpatrick M, Darzi A, Birnbach DJ. "Priming" hand hygiene compliance in clinical environments. Health Psychol. 2016 Jan;35(1):96-101. doi: 10.1037/hea0000239. Epub 2015 Jul 27. PMID 26214075
- [Derived] Gilmartin H, Saint S, Rogers M, Winter S, Snyder A, Quinn M, Chopra V. Pilot randomised controlled trial to improve hand hygiene through mindful moments. BMJ Qual Saf. 2018 Oct;27(10):799-806. doi: 10.1136/bmjqs-2017-007359. Epub 2018 Feb 20. PMID 29463769